CLINICAL TRIAL: NCT05790356
Title: Fecal Microbial Transplantation for Rheumatoid Arthritis Trial
Acronym: FeMiTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FeMiTRA01
Record Dates: First submitted 2023-02-15; First posted 2023-03-30 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Arthritis; Arthritis, Rheumatoid; Fecal Microbiota Transplantation
Keywords: Arthritis; Rheumatoid; Rheumatoid Arthritis; clinical trial; fecal matter transplantation; fecal matter transplant; faecal; autoimmune; proof of concept
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled proof-of-concept study.
Who Masked: Participant, Investigator
Masking Description: Neither the participants or the investigator will know which treatment arms participants have been assigned to. This information can be obtained quickly from pharmacy if needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbial Transplant (Experimental): Participants will be administered 35-40 FMT capsules orally with water, for a total dose of 80-100g. This will only occur once and takes approximately 30 minutes.
  Interventions: Drug: Fecal Microbial transplant
- Placebo (Placebo Comparator): Participants will be administered 35-40 placebo capsules orally with water. This will only occur once and takes approximately 30 minutes.
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Drug: Fecal Microbial transplant — Fecal microbial transplant will be investigated for its effect on gut bacterial composition in patients with rheumatoid arthritis.
  Other Names: FMT Capsules
  Arms: Fecal Microbial Transplant
Other: Placebo capsules — The placebo capsules will not contain FMT but will have the same appearance.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This clinical trial will investigate the effects of capsules containing stool from healthy donors, called fecal microbial transplant (FMT), in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled proof-of-concept trial. A total of 30 RA patients will be asked to join the study. They will be randomized to receive capsular FMT + standard of care or placebo + standard of care. There will be four study visits in total: Baseline, FMT administration, 6- and 12-week follow-up visits. Follow-up visits will consist of assessment by a rheumatologist, completion of surveys, and collection of biologic samples.

Samples for the study are stool, urine and blood. Blood and fecal samples will be collected at baseline, 6 weeks and 12 weeks. Urine samples will be collected at baseline and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-years old or older
* RA diagnosis by ACR/EULAR criteria [26]
* Positive for the RA-associated antibodies, anti-citrullinated protein/peptide antibodies (ACPA) and/or rheumatoid factor (RF)
* Stable RA therapy > 6 months
* Patient in remission or low disease activity by DAS28
* Consents to study

Fecal Donor Inclusion Criteria:

* A healthy donor who has a normal body mass index (BMI of 18.5-30) and who satisfies the following criteria will be selected from a pool of donors available in the Infectious Diseases clinic at St. Joseph's Hospital supervised by Dr. Silverman and screened for all transmissible agents. at the Microbiology and Immunology lab at St. Joseph's Hospital under Dr. Silverman for the study and screened for transmissible agents.

Exclusion Criteria:

* Pregnant or breastfeeding
* Current or recent [in the last 60 days] exposure to high dose oral (>30 mg of prednisone daily or equivalent), IV corticosteroids, biologic therapies or JAKi.
* Patients who require inhaled steroids or local steroid injections are not excluded from the study
* Has a diagnosis of immunodeficiency (HIV, transplantation, or autoimmune disease other than RA requiring immunosuppressive therapies), or currently receiving systemic steroid therapy (>10 mg prednisone daily or equivalent)
* Received rituximab or other chemotherapeutic agent in the last 2 years.
* Expected to require any other form of systemic or localized anti-neoplastic therapy while on study
* Has a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the patient has undergone potentially curative therapy with no evidence of that disease for five years. NOTE: This time requirement also does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers.
* Ongoing use of antibiotics/anti-virals or previous use of antibiotics/anti-virals in the last 3 months prior to the FMT procedure
* Has an active infection requiring systemic therapy or requiring hospital admission in last 3 months.
* Presence of a chronic intestinal disease (e.g. Celiac disease, malabsorption, colonic tumor, IBD)
* Presence of absolute contra-indications to FMT administration
* Toxic megacolon
* Anaphylactic allergic reactions to food (e.g. shellfish, nuts, seafood, eggs)
* Has serious uncontrolled concomitant illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), severe obstructive or restrictive pulmonary diseases, cirrhosis or ALT>100, renal disease with GFR<50 and uncontrolled psychiatric illness.
* Patient has received a live vaccine within 4 weeks prior to the first dose of treatment
* Insulin-dependent diabetes
* Previous bariatric surgery
* Chronic neutropenia (<0.5) Currently participating in another clinical trial

Fecal Donor Exclusion Criteria:

* Any underlying metabolic disease including; hypertension, hyperlipidemia, diabetes, insulin insensitivity, atherosclerosis
* A history of any gastrointestinal or liver disorders or cancers. Including but not limited to; gastroesophageal reflux, peptic ulcer disease, celiac disease, inflammatory bowel disease (Crohn's disease or ulcerative colitis), microscopic colitis, motility disorders (including gastroparesis and irritable bowel syndrome) diverticular disease
* Previous surgery to the intestine, liver or gallbladder (except remote appendectomy)
* History of any malignancy
* Use within 3 months of any antibiotics
* Hospitalization within 3 months
* Recent travel to a developing country (within 3 months).
* New Sexual Partner (within 3 months)
* Street drug use, family history of diabetes, early onset coronary disease or gastrointestinal or liver disease, colon cancer, familial malignancy
* Psychiatric history (major affective disorder, psychotic illness, ongoing use of any psychiatric medications)
* Any positive laboratory results for a transmissible pathogen
* Alcohol intake with a cut off value of <10g/d in women and <20g/d in men
* Currently participating in another clinical trial that may alter fecal composition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Intestinal Permeability | Baseline and 6 weeks
  A blood sample will be collected for bacterial DNA analysis.
Change in Intestinal Permeability | Baseline and 6 weeks
  A urine sample will be collected to measure the lactulose to mannitol ratio.
Change in RA-associated autoantibodies | Baseline, 6 weeks and 12 weeks
  A blood sample will be collected to measure RA-associated autoantibodies.
Adverse Events | Baseline
  Adverse events will be evaluated at every study visit. Participants will also be instructed to contact study staff by phone if they experience an adverse event in between study visits.
Adverse Events | FMT treatment visit
  Adverse events will be evaluated at every study visit. Participants will also be instructed to contact study staff by phone if they experience an adverse event in between study visits.
Adverse Events | 6 weeks post-treatment
  Adverse events will be evaluated at every study visit. Participants will also be instructed to contact study staff by phone if they experience an adverse event in between study visits.
Adverse Events | 12 weeks post-treatment
  Adverse events will be evaluated at every study visit. Participants will also be instructed to contact study staff by phone if they experience an adverse event in between study visits.

SECONDARY OUTCOMES:
Change in Fecal Microbial Composition | Baseline, 6 weeks and 12 weeks
  Stool samples will be collected to determine fecal microbial composition using 16S-RNA sequencing.
Change in C-Reactive Protein | Baseline, 6 weeks and 12 weeks.
  Blood sample will be collected to measure CRP levels.

OTHER OUTCOMES:
Pain Visual Analog Scale | Baseline, 6 weeks and 12 weeks
  Change in pain will be measured using a visual analog scale.
Fatigue | Baseline, 6 weeks and 12 weeks
  Change in fatigue will be measured with a visual analog scale.
Sleep | Baseline, 6 weeks and 12 weeks
  Change in sleep will be measured with a visual analog scale.
Change in RA disease activity | Baseline, 6 weeks and 12 weeks
  RA disease activity will be measured using the disease activity score-28 (DAS28).
Change in RA disease activity | Baseline, 6 weeks and 12 weeks
  RA disease activity will be measured using the health assessment questionnaire (HAQ).
Change in RA disease activity | Baseline, 6 weeks and 12 weeks
  RA disease activity will be measured using the clinical disease activity index (CDAI).
Insulin Resistance | Baseline, 6 weeks and 12 weeks
  Fasting glucose and insulin will be measured from a blood sample to calculate the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Blood Pressure | Baseline, 6 weeks and 12 weeks
  Systolic and Diastolic blood pressure is part of the standard of care and will be measured at each study visit.
Body Mass Index | Baseline, 6 weeks and 12 weeks
  Body mass index is part of the standard of care and will be measured at each study visit.
Patient Acceptability of FMT | Baseline, 6 weeks and 12 weeks
  Participants will complete an acceptability of therapy survey for FMT. The survey asks them questions about how well the FMT process was explained to them, and how they feel about it. The participant is asked to select one answer per question ranging from :strongly agree" to "strongly disagree"
Tolerability of DMARD Therapy | Baseline, 6 weeks and 12 weeks
  Participants will complete a survey on tolerability of DMARD therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Barra, MD, MPH, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

REFERENCES:
- [Background] Bykerk VP, Akhavan P, Hazlewood GS, Schieir O, Dooley A, Haraoui B, Khraishi M, Leclercq SA, Legare J, Mosher DP, Pencharz J, Pope JE, Thomson J, Thorne C, Zummer M, Bombardier C; Canadian Rheumatology Association. Canadian Rheumatology Association recommendations for pharmacological management of rheumatoid arthritis with traditional and biologic disease-modifying antirheumatic drugs. J Rheumatol. 2012 Aug;39(8):1559-82. doi: 10.3899/jrheum.110207. Epub 2011 Sep 15. PMID 21921096
- [Background] Barnabe C, Sun Y, Boire G, Hitchon CA, Haraoui B, Thorne JC, Tin D, van der Heijde D, Curtis JR, Jamal S, Pope JE, Keystone EC, Bartlett S, Bykerk VP; CATCH Investigators. Heterogeneous Disease Trajectories Explain Variable Radiographic, Function and Quality of Life Outcomes in the Canadian Early Arthritis Cohort (CATCH). PLoS One. 2015 Aug 24;10(8):e0135327. doi: 10.1371/journal.pone.0135327. eCollection 2015. PMID 26301589
- [Background] Bombardier C, Hazlewood GS, Akhavan P, Schieir O, Dooley A, Haraoui B, Khraishi M, Leclercq SA, Legare J, Mosher DP, Pencharz J, Pope JE, Thomson J, Thorne C, Zummer M, Gardam MA, Askling J, Bykerk V; Canadian Rheumatology Association. Canadian Rheumatology Association recommendations for the pharmacological management of rheumatoid arthritis with traditional and biologic disease-modifying antirheumatic drugs: part II safety. J Rheumatol. 2012 Aug;39(8):1583-602. doi: 10.3899/jrheum.120165. Epub 2012 Jun 15. PMID 22707613
- [Background] Munro S, Spooner L, Milbers K, Hudson M, Koehn C, Harrison M. Perspectives of patients, first-degree relatives and rheumatologists on preventive treatments for rheumatoid arthritis: a qualitative analysis. BMC Rheumatol. 2018 Jul 5;2:18. doi: 10.1186/s41927-018-0026-7. eCollection 2018. PMID 30886969
- [Background] Loyola-Sanchez A, Hazlewood G, Crowshoe L, Linkert T, Hull PM, Marshall D, Barnabe C. Qualitative Study of Treatment Preferences for Rheumatoid Arthritis and Pharmacotherapy Acceptance: Indigenous Patient Perspectives. Arthritis Care Res (Hoboken). 2020 Apr;72(4):544-552. doi: 10.1002/acr.23869. PMID 30821924
- [Background] Taylor PC, Ancuta C, Nagy O, de la Vega MC, Gordeev A, Jankova R, Kalyoncu U, Lagunes-Galindo I, Morovic-Vergles J, de Souza MPGUES, Rojkovich B, Sidiropoulos P, Kawakami A. Treatment Satisfaction, Patient Preferences, and the Impact of Suboptimal Disease Control in a Large International Rheumatoid Arthritis Cohort: SENSE Study. Patient Prefer Adherence. 2021 Feb 17;15:359-373. doi: 10.2147/PPA.S289692. eCollection 2021. PMID 33633444
- [Background] Deane KD, Holers VM. Rheumatoid Arthritis Pathogenesis, Prediction, and Prevention: An Emerging Paradigm Shift. Arthritis Rheumatol. 2021 Feb;73(2):181-193. doi: 10.1002/art.41417. Epub 2020 Dec 8. PMID 32602263
- [Background] Wilson AS, Koller KR, Ramaboli MC, Nesengani LT, Ocvirk S, Chen C, Flanagan CA, Sapp FR, Merritt ZT, Bhatti F, Thomas TK, O'Keefe SJD. Diet and the Human Gut Microbiome: An International Review. Dig Dis Sci. 2020 Mar;65(3):723-740. doi: 10.1007/s10620-020-06112-w. PMID 32060812
- [Background] Zaiss MM, Joyce Wu HJ, Mauro D, Schett G, Ciccia F. The gut-joint axis in rheumatoid arthritis. Nat Rev Rheumatol. 2021 Apr;17(4):224-237. doi: 10.1038/s41584-021-00585-3. Epub 2021 Mar 5. PMID 33674813
- [Background] Scher JU, Sczesnak A, Longman RS, Segata N, Ubeda C, Bielski C, Rostron T, Cerundolo V, Pamer EG, Abramson SB, Huttenhower C, Littman DR. Expansion of intestinal Prevotella copri correlates with enhanced susceptibility to arthritis. Elife. 2013 Nov 5;2:e01202. doi: 10.7554/eLife.01202. PMID 24192039
- [Background] Mohammed AT, Khattab M, Ahmed AM, Turk T, Sakr N, M Khalil A, Abdelhalim M, Sawaf B, Hirayama K, Huy NT. The therapeutic effect of probiotics on rheumatoid arthritis: a systematic review and meta-analysis of randomized control trials. Clin Rheumatol. 2017 Dec;36(12):2697-2707. doi: 10.1007/s10067-017-3814-3. Epub 2017 Sep 15. PMID 28914373
- [Background] Meyers S, Shih J, Neher JO, Safranek S. Clinical Inquiries: How effective and safe is fecal microbial transplant in preventing C difficile recurrence? J Fam Pract. 2018 Jun;67(6):386-388. PMID 29879241
- [Background] Claytor JD, El-Nachef N. Fecal microbial transplant for inflammatory bowel disease. Curr Opin Clin Nutr Metab Care. 2020 Sep;23(5):355-360. doi: 10.1097/MCO.0000000000000676. PMID 32618725
- [Background] Chapman BC, Moore HB, Overbey DM, Morton AP, Harnke B, Gerich ME, Vogel JD. Fecal microbiota transplant in patients with Clostridium difficile infection: A systematic review. J Trauma Acute Care Surg. 2016 Oct;81(4):756-64. doi: 10.1097/TA.0000000000001195. PMID 27648772
- [Background] Sun D, Li W, Li S, Cen Y, Xu Q, Li Y, Sun Y, Qi Y, Lin Y, Yang T, Xu P, Lu Q. Fecal Microbiota Transplantation as a Novel Therapy for Ulcerative Colitis: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2016 Jun;95(23):e3765. doi: 10.1097/MD.0000000000003765. PMID 27281075
- [Background] Kao D, Roach B, Silva M, Beck P, Rioux K, Kaplan GG, Chang HJ, Coward S, Goodman KJ, Xu H, Madsen K, Mason A, Wong GK, Jovel J, Patterson J, Louie T. Effect of Oral Capsule- vs Colonoscopy-Delivered Fecal Microbiota Transplantation on Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2017 Nov 28;318(20):1985-1993. doi: 10.1001/jama.2017.17077. PMID 29183074
- [Background] Wang S, Xu M, Wang W, Cao X, Piao M, Khan S, Yan F, Cao H, Wang B. Systematic Review: Adverse Events of Fecal Microbiota Transplantation. PLoS One. 2016 Aug 16;11(8):e0161174. doi: 10.1371/journal.pone.0161174. eCollection 2016. PMID 27529553
- [Background] Craven LJ, Nair Parvathy S, Tat-Ko J, Burton JP, Silverman MS. Extended Screening Costs Associated With Selecting Donors for Fecal Microbiota Transplantation for Treatment of Metabolic Syndrome-Associated Diseases. Open Forum Infect Dis. 2017 Nov 6;4(4):ofx243. doi: 10.1093/ofid/ofx243. eCollection 2017 Fall. PMID 29255739
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Vehreschild MJ, Cornely OA. Fecal Microbiota Transfer 2.0. J Infect Dis. 2016 Jul 15;214(2):169-70. doi: 10.1093/infdis/jiv768. Epub 2016 Feb 8. No abstract available. PMID 26908719
- [Background] Neill J, Belan I, Ried K. Effectiveness of non-pharmacological interventions for fatigue in adults with multiple sclerosis, rheumatoid arthritis, or systemic lupus erythematosus: a systematic review. J Adv Nurs. 2006 Dec;56(6):617-35. doi: 10.1111/j.1365-2648.2006.04054.x. PMID 17118041
- [Background] Gwinnutt JM, Wieczorek M, Balanescu A, Bischoff-Ferrari HA, Boonen A, Cavalli G, de Souza S, de Thurah A, Dorner TE, Moe RH, Putrik P, Rodriguez-Carrio J, Silva-Fernandez L, Stamm T, Walker-Bone K, Welling J, Zlatkovic-Svenda MI, Guillemin F, Verstappen SMM. 2021 EULAR recommendations regarding lifestyle behaviours and work participation to prevent progression of rheumatic and musculoskeletal diseases. Ann Rheum Dis. 2023 Jan;82(1):48-56. doi: 10.1136/annrheumdis-2021-222020. Epub 2022 Mar 8. PMID 35260387
- [Background] Skoldstam L, Hagfors L, Johansson G. An experimental study of a Mediterranean diet intervention for patients with rheumatoid arthritis. Ann Rheum Dis. 2003 Mar;62(3):208-14. doi: 10.1136/ard.62.3.208. PMID 12594104
- [Background] Holers VM, Demoruelle MK, Kuhn KA, Buckner JH, Robinson WH, Okamoto Y, Norris JM, Deane KD. Rheumatoid arthritis and the mucosal origins hypothesis: protection turns to destruction. Nat Rev Rheumatol. 2018 Sep;14(9):542-557. doi: 10.1038/s41584-018-0070-0. PMID 30111803
- [Background] Svard A, Roos Ljungberg K, Brink M, Martinsson K, Sjowall C, Rantapaa Dahlqvist S, Kastbom A. Secretory antibodies to citrullinated peptides in plasma and saliva from rheumatoid arthritis patients and their unaffected first-degree relatives. Clin Exp Immunol. 2020 Feb;199(2):143-149. doi: 10.1111/cei.13381. Epub 2019 Oct 22. PMID 31605388
- [Background] Kay J, Upchurch KS. ACR/EULAR 2010 rheumatoid arthritis classification criteria. Rheumatology (Oxford). 2012 Dec;51 Suppl 6:vi5-9. doi: 10.1093/rheumatology/kes279. PMID 23221588
- [Background] Craven L, Rahman A, Nair Parvathy S, Beaton M, Silverman J, Qumosani K, Hramiak I, Hegele R, Joy T, Meddings J, Urquhart B, Harvie R, McKenzie C, Summers K, Reid G, Burton JP, Silverman M. Allogenic Fecal Microbiota Transplantation in Patients With Nonalcoholic Fatty Liver Disease Improves Abnormal Small Intestinal Permeability: A Randomized Control Trial. Am J Gastroenterol. 2020 Jul;115(7):1055-1065. doi: 10.14309/ajg.0000000000000661. PMID 32618656
- [Background] Al KF, Bisanz JE, Gloor GB, Reid G, Burton JP. Evaluation of sampling and storage procedures on preserving the community structure of stool microbiota: A simple at-home toilet-paper collection method. J Microbiol Methods. 2018 Jan;144:117-121. doi: 10.1016/j.mimet.2017.11.014. Epub 2017 Nov 16. PMID 29155236
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Aletaha D, Ward MM, Machold KP, Nell VP, Stamm T, Smolen JS. Remission and active disease in rheumatoid arthritis: defining criteria for disease activity states. Arthritis Rheum. 2005 Sep;52(9):2625-36. doi: 10.1002/art.21235. PMID 16142705
- [Background] Daisley BA, Chanyi RM, Abdur-Rashid K, Al KF, Gibbons S, Chmiel JA, Wilcox H, Reid G, Anderson A, Dewar M, Nair SM, Chin J, Burton JP. Abiraterone acetate preferentially enriches for the gut commensal Akkermansia muciniphila in castrate-resistant prostate cancer patients. Nat Commun. 2020 Sep 24;11(1):4822. doi: 10.1038/s41467-020-18649-5. PMID 32973149